CLINICAL TRIAL: NCT00994318
Title: An Open-label, Multicentre, Randomised, 3-arm Study to Investigate the Comparative Efficacy and Safety of Intravenous Ferric Carboxymaltose (Ferinject High and Low Dosage Regimens) Versus Oral Iron for the Treatment of Iron Deficiency Anaemia in Subjects With Non-dialysis-dependent Chronic Kidney Disease
Brief Title: Ferric Carboxymaltose (FCM) Assessment in Subjects With Iron Deficiency Anaemia and Non-dialysis-dependent Chronic Kidney Disease (NDD-CKD)
Acronym: FIND-CKD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vifor Pharma (Industry)
Collaborators: American Regent, Inc. (Industry); ICON Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FER-CKD-01
Record Dates: First submitted 2009-10-12; First posted 2009-10-14 (Estimated); Results first posted 2014-05-07 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Iron Deficiency Anaemia; Chronic Kidney Disease
Keywords: Ferinject Iron Deficiency Anaemia Chronic Kidney Disease
MeSH Terms: conditions — Anemia, Iron-Deficiency; Renal Insufficiency, Chronic | interventions — Fosfomycin; ferric carboxymaltose; Iron; ferrous sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- FCM (high ferritin target) (Experimental): Ferric carboxymaltose (FCM) (Ferinject / Injectafer) targeting ferritin level of 400 - 600 mcg/L
  Interventions: Drug: FCM (Ferric carboxymaltose) high ferritin target
- FCM (low ferritin target) (Experimental): Ferric carboxymaltose (FCM) (Ferinject / Injectafer) targeting ferritin level of 100 - 200 mcg/L
  Interventions: Drug: FCM (Ferric carboxymaltose) low ferritin target
- Oral Iron (Active Comparator): Ferrous sulphate 100 mg iron twice daily, continuous
  Interventions: Drug: Oral Iron (Ferrous sulphate)

INTERVENTIONS:
Drug: FCM (Ferric carboxymaltose) high ferritin target
  Other Names: Ferinject; Injectafer
  Arms: FCM (high ferritin target)
Drug: FCM (Ferric carboxymaltose) low ferritin target
  Other Names: Ferinject; Injectafer
  Arms: FCM (low ferritin target)
Drug: Oral Iron (Ferrous sulphate)
  Other Names: Ferrous sulphate
  Arms: Oral Iron

SUMMARY:
Phase IIIb study to evaluate the long-term efficacy of ferric carboxymaltose (FCM) (using targeted ferritin levels to determine dosing) or oral iron in non-dialysis-dependent chronic kidney disease (NDD-CKD) subjects with iron deficiency anaemia (IDA).

DETAILED DESCRIPTION:
After an initial screening period of up to 4 weeks, eligible subjects were randomised (1:1:2) to 1 of the following 3 treatment arms for a period of 52 weeks.

1. FCM regimen (maximum single intravenous doses of 1,000 mg of iron) targeting a ferritin level of 400-600 mcg/L.
2. FCM regimen (maximum single intravenous doses of 200 mg of iron) targeting a ferritin level of 100-200 mcg/L.
3. Daily oral iron with 200 mg iron/day (100 mg twice daily)

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age.
2. NDD-CKD subjects with an estimated glomerular filtration rate (eGFR) ≤60 mL/min/1.73 m2 using modification of diet in renal disease 4 (MDRD-4) calculation.
3. NDD-CKD subjects with an eGFR loss ≤12 mL/min/1.73 m2/year and a predicted eGFR of ≥15 mL/min/1.73 m2 in 12 months.
4. Any single Hb between 9 and 11 g/dL within 4 weeks of randomisation. A value taken as part of routine medical care was used.
5. Any single serum ferritin <100 mcg/L or <200 mcg/L with TSAT <20% within 4 weeks of randomisation. Measurements taken as part of routine medical care were used.
6. ESA naïve; no exposure to ESA in last 4 months prior to randomisation.
7. Females of childbearing potential must have had a negative pregnancy test, using any medically acceptable assessment, prior to randomisation.
8. Before any study specific procedure, the appropriate written informed consent must have been obtained.

Exclusion Criteria:

1. History of acquired iron overload.
2. Known hypersensitivity reaction to any component of ferrous sulphate or FCM. Subjects with hypersensitivity to other forms of iron were permitted to participate.
3. Documented history of discontinuing oral iron products due to significant gastrointestinal (GI) distress.
4. Screening TSAT >40%.
5. Known active infection, C-reactive protein >20 mg/L, clinically significant overt bleeding, active malignancy (i.e., clinical evidence of current malignancy or not in stable remission for at least 5 years since completion of last treatment with exception of basal cell or squamous cell carcinoma of the skin, and cervical intraepithelial neoplasia).
6. History of chronic alcohol abuse (alcohol consumption >40 g/day).
7. Chronic liver disease and/or screening alanine transaminase or aspartate transaminase above 3 times the upper limit of the normal range.
8. Active human immunodeficiency virus (HIV)/acquired immunodeficiency syndrome or active hepatitis B or C virus infection.
9. Anaemia due to reasons other than iron deficiency (e.g., haemoglobinopathy). Subjects with treated Vitamin B12 or folic acid deficiency were permitted.
10. IV iron and/or blood transfusion in previous 30 days prior to screening (or during the screening period).
11. Oral iron therapy at doses >100 mg/day dosing must have been discontinued at least 1 week prior to randomisation. If subject had received this therapy for >3 months (at doses >100 mg/day) then subject was not eligible. Ongoing use of multivitamins containing iron was permitted.
12. Immunosuppressive therapy that may have led to anaemia (e.g., cyclophosphamide, azathioprine, or mycophenolate mofetil). Steroid therapy was permitted.
13. Currently requiring renal dialysis.
14. Anticipated dialysis or transplant during the study.
15. Anticipated need for surgery that may have resulted in significant bleeding (>100 mL).
16. Currently suffering from chronic heart failure New York Heart Association Class IV.
17. Poorly controlled hypertension (>160 mmHg systolic pressure or >100 mmHg diastolic pressure).
18. Acute coronary syndrome or stroke within the 3 months prior to screening.
19. Currently suffering from concomitant, severe psychiatric disorders or other conditions which, in the opinion of the Investigator, would have made participation unacceptable.
20. Subject was not using adequate contraceptive precautions.
21. Subject of childbearing potential was evidently pregnant (e.g., positive human chorionic gonadotropin test) or was breast feeding.
22. Body weight <35 kg.
23. Subject currently was enrolled in or had not yet completed at least 30 days since ending other investigational device or drug studies, or subject was receiving other investigational agent(s).
24. Subject would not be available for follow-up assessment.
25. Subject had any kind of disorder that compromised the ability of the subject to give written informed consent and/or to comply with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 626 (Actual)
Dates: Start 2009-12; Primary Completion 2013-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Iain Macdougall, Principal Investigator — King's College Hospital NHS Trust
Locations (19):
- Trial Management Associates, Wilmington, North Carolina, United States
- Gosford Hospital - Renal Research, Gosford, Australia
- Medizinische Universität Innsbruck Univ.-Klinik für Innere Medizin IV, Innsbruck, Austria
- RHMS Baudour - Department of Nephrology and Dialysis, Baudour, Belgium
- Nemocnice s poliklinikou v Novem Jicine, p.o. p.o. Interni oddeleni - nefrologie a dialyza, Nový Jičín, Czechia
- Lillebalt Frederica Sygehus Department of Nephrology, Frederica, Denmark
- CHU grenoble - Service de Nephrologie, Grenoble, France
- Praxis Dr. Kraatz, Demmin, Germany
- General Hospital of Arta - Nephrology Department, Arta, Greece
- Ospedali Riuniti Anzio-Nettuno ASL ROMA H U.O. Nefrologia e Dialisi, Anzio, Italy
- Meander Medisch Centrum - Locatie Amersfoort Lichtenberg, Amersfoort, Netherlands
- St. Olav's Hospital, Trondheim, Norway
- Miedzyleski Szpital Spec. Oddzial I Wewnetrzny I Nefrologii, Warsaw, Poland
- Hospital Santa Maria - Nefrologia, Lisbon, Portugal
- Spitalul Clinic de Nefrologie"Dr Carol Davila", Bucharest, Romania
- Hospital Universitario Marqués de Valdecilla - Servicio de Nefrología, Santander, Spain
- Karolinska University Hospital, Stockholm, Sweden
- Cukurova University Medical Faculty Balcali Hospital - Department of Nephrology, Adana, Turkey (Türkiye)
- King's College Hospital, London, United Kingdom

REFERENCES:
- [Derived] Roger SD, Gaillard CA, Bock AH, Carrera F, Eckardt KU, Van Wyck DB, Cronin M, Meier Y, Larroque S, Macdougall IC; FIND-CKD Study Investigators. Safety of intravenous ferric carboxymaltose versus oral iron in patients with nondialysis-dependent CKD: an analysis of the 1-year FIND-CKD trial. Nephrol Dial Transplant. 2017 Sep 1;32(9):1530-1539. doi: 10.1093/ndt/gfw264. PMID 28339831
- [Derived] Macdougall IC, Bock AH, Carrera F, Eckardt KU, Gaillard C, Van Wyck D, Meier Y, Larroque S, Roger SD; FIND-CKD Study investigators. Renal function in patients with non-dialysis chronic kidney disease receiving intravenous ferric carboxymaltose: an analysis of the randomized FIND-CKD trial. BMC Nephrol. 2017 Jan 17;18(1):24. doi: 10.1186/s12882-017-0444-6. PMID 28095881
- [Derived] Macdougall IC, Bock AH, Carrera F, Eckardt KU, Gaillard C, Van Wyck D, Roubert B, Nolen JG, Roger SD; FIND-CKD Study Investigators. FIND-CKD: a randomized trial of intravenous ferric carboxymaltose versus oral iron in patients with chronic kidney disease and iron deficiency anaemia. Nephrol Dial Transplant. 2014 Nov;29(11):2075-84. doi: 10.1093/ndt/gfu201. Epub 2014 Jun 2. PMID 24891437

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | FCM (High Ferritin Target) | FCM (Low Ferritin Target) | Oral Iron
Started | 155 | 154 | 317
Completed | 133 | 136 | 250
Not Completed | 22 | 18 | 67

BASELINE CHARACTERISTICS:
Population: Baseline analysis population is the Full Analysis Set (FAS); all subjects randomised to treatment, received at least 1 dose study drug or, per protocol, not treated due to ferritin <100 mcg/L, and attended at least 1 post-baseline visit with at least 1 non-missing assessment. Overall 626 subjects were randomised, the FAS consists of 613 subjects.
Groups:
- FCM (High Ferritin Target: Ferric carboxymaltose (FCM) (Ferinject / Injectafer) targeting ferritin level of 400 - 600 mcg/L
- Total: Total of all reporting groups
Arm/Group | FCM (High Ferritin Target | FCM (Low Ferritin Target) | Oral Iron | Total
Number analyzed (Participants) | 153 | 152 | 308 | 613
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 41 | 49 | 92 | 182
  >=65 years | 112 | 103 | 216 | 431
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.46 (12.643) | 68.19 (13.264) | 69.31 (13.404) | 69.07 (13.172)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 98 | 192 | 381
  Male | 62 | 54 | 116 | 232
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 3 | 9 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 2 | 5 | 7 | 14
  White | 149 | 144 | 291 | 584
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 7 | 14
  Portugal | 2 | 2 | 5 | 9
  Greece | 28 | 28 | 55 | 111
  Turkey | 7 | 7 | 15 | 29
  Austria | 2 | 2 | 4 | 8
  United Kingdom | 17 | 18 | 36 | 71
  Italy | 10 | 10 | 19 | 39
  France | 1 | 0 | 3 | 4
  Czech Republic | 16 | 15 | 31 | 62
  Belgium | 3 | 3 | 4 | 10
  Poland | 11 | 11 | 20 | 42
  Romania | 2 | 2 | 4 | 8
  Australia | 15 | 16 | 31 | 62
  Denmark | 1 | 1 | 2 | 4
  Germany | 26 | 25 | 49 | 100
  Netherlands | 4 | 4 | 8 | 16
  Norway | 0 | 1 | 4 | 5
  Sweden | 0 | 0 | 1 | 1
  Spain | 4 | 4 | 10 | 18

OUTCOME MEASURES:

1. Primary Outcome: Kaplan-Meier Survival Analysis for Time to Other Anemia Therapy or Hb Trigger
Description: Endpoint reported number of participants with/without events and was reached:
  * First time of initiation of additional or alternative anaemia management,
  * First time the subject reached the Hb trigger.
    3 primary comparisons using a hierarchical step-down procedure on the log-rank test to preserve an alpha level of 0.05, performed in the following order:
    1. FCM (high ferritin target) compared with oral iron.
    2. FCM (high ferritin target) compared with FCM (low ferritin target).
    3. FCM (low ferritin target) compared with oral iron.
  Sensitivity analyses of the primary endpoint were performed using the following alternative definitions of time to initiation of additional or alternative anaemia management:
  1. Without taking into account the Hb trigger.
  2. Taking into account the Hb trigger based on local laboratory data, instead of central laboratory data.
  3. Taking into account the Hb trigger based on subjects with a complete set of Hb values from the central laboratory.
Time Frame: Up to 1 year after baseline
Population: The Full Analysis Set (FAS) was used for the primary endpoint analysis, which consisted of all subjects randomised to treatment, received at least 1 dose of study treatment or, according to the protocol, were not treated due to ferritin value <100 mcg/L, and attended at least 1 post-baseline visit with at least 1 non-missing assessment available.
Measure: Number; unit: participants
Groups:
- FCM (High Ferritin Target): Ferric carboxymaltose (FCM) (Ferinject / Injectafer), targeting ferritin level of 400-600 mcg/L
- FCM (Low Ferritin Level): Ferric carboxymaltose (FCM) (Ferinject / Injectafer), targeting ferritin level of 100-200 mcg/L
Arm/Group | FCM (High Ferritin Target) | FCM (Low Ferritin Level) | Oral Iron
Number analyzed (Participants) | 153 | 152 | 308
participants
  Number of patients with events | 36 (7.65) | 49 (9.47) [0.45 to 1.05] | 98 (7.71) [0.44 to 0.95]
  Number of patients without events | 117 | 103 | 210
Statistical Analysis 1: Comparison: FCM (High Ferritin Target) vs Oral Iron; FCM (Ferinject / Injectafer) targeting high ferritin level (400 - 600 mcg/L) compared with Oral Iron (Ferrous sulphate 100 mg iron twice daily). Three primary comparisons using a hierarchical step-down procedure on the log-rank test to preserve the overall alpha level of 0.05, performed in the following order: 1. FCM (high ferritin target) compared with oral iron. 2. FCM (high ferritin target) compared with FCM (low ferritin target). 3. FCM (low ferritin target) compared with oral iron; Test type: Superiority or Other; p = 0.026, Log Rank; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.44 to 0.95]
Statistical Analysis 2: Comparison: FCM (High Ferritin Target) vs FCM (Low Ferritin Level); FCM (Ferinject / Injectafer) targeting high ferritin level (400-600mcg/L) compared with FCM targeting low ferritin level (100 - 200 mcg/L). Three primary comparisons using a hierarchical step-down procedure on the log-rank test to preserve the overall alpha level of 0.05, performed in the following order: 1. FCM (high ferritin target) compared with oral iron. 2. FCM (high ferritin target) compared with FCM (low ferritin target). 3. FCM (low ferritin target) compared with oral iron; Test type: Superiority or Other; p = 0.082, Log Rank; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.45 to 1.05]
Statistical Analysis 3: Comparison: FCM (High Ferritin Target) vs Oral Iron; Sensitivity analysis of the primary endpoint. Time to initiation of additional or alternative anaemia management without taking into account the Hb trigger. FCM (Ferinject / Injectafer) targeting high ferritin level (400 - 600 mcg/L) compared with Oral Iron (Ferrous sulphate 100 mg iron twice daily); Test type: Superiority or Other; p = 0.020, Log Rank; Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.39 to 0.93]
Statistical Analysis 4: Comparison: FCM (High Ferritin Target) vs FCM (Low Ferritin Level); Sensitivity analysis of the primary endpoint. Time to initiation of additional or alternative anaemia management taking into account the Hb trigger based on local laboratory data, instead of central laboratory data. FCM (Ferinject / Injectafer) targeting high ferritin level (400 - 600 mcg/L) compared with Oral Iron (Ferrous sulphate 100 mg iron twice daily); Test type: Superiority or Other; p = 0.008, Log Rank; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.43 to 0.88]
Statistical Analysis 5: Comparison: FCM (High Ferritin Target) vs Oral Iron; Sensitivity analysis of the primary endpoint. Time to initiation of additional or alternative anaemia management taking into account the Hb trigger based on subjects with a complete set of Hb values from central laboratory. FCM (Ferinject / Injectafer) targeting high ferritin level (400 - 600 mcg/L) compared with Oral Iron (Ferrous sulphate 100 mg iron twice daily); Test type: Superiority or Other; p = 0.12, Log Rank; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.45 to 1.10]

ADVERSE EVENTS:
Time Frame: Adverse Event data was collected for 56 weeks after baseline.
Description: The Number of Patients at Risk is the Safety Set which consists of all randomised subjects who received at least 1 dose of study drug.
Arm/Group | FCM (High Ferritin Target) | FCM (Low Ferritin Target) | Oral Iron
Serious Adverse Events (participants affected / at risk) | 39/154 | 36/150 | 59/312
Other Adverse Events (participants affected / at risk) | 126/154 | 129/150 | 255/312
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FCM (High Ferritin Target) (N=154) | FCM (Low Ferritin Target) (N=150) | Oral Iron (N=312)
Acute Myocardial Infarction (Cardiac disorders) | 2 | 0 | 4
Cardiac Failure (Cardiac disorders) | 1 | 0 | 3
Cardiac Failure Congestive (Cardiac disorders) | 2 | 1 | 1
Acute Coronary Syndrome (Cardiac disorders) | 2 | 0 | 1
Myocardial Infarction (Cardiac disorders) | 1 | 1 | 1
Cardiac Arrest (Cardiac disorders) | 1 | 0 | 1
Coronary Artery Disease (Cardiac disorders) | 0 | 1 | 1
Angina Unstable (Cardiac disorders) | 0 | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 0 | 0
Atrioventricular Block Complete (Cardiac disorders) | 0 | 0 | 1
Cardiac Failure Acute (Cardiac disorders) | 0 | 1 | 0
Extrasystoles (Cardiac disorders) | 0 | 0 | 1
Hypertensive Heart Disease (Cardiac disorders) | 0 | 0 | 1
Left Ventricular Dysfunction (Cardiac disorders) | 1 | 0 | 0
Myocardial Ischaemia (Cardiac disorders) | 0 | 1 | 0
Sinus Arrhythmia (Cardiac disorders) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 4
Urinary Tract Infection (Infections and infestations) | 1 | 0 | 2
Infective Exacerbation of Chronic Obstructive Airways Disease (Infections and infestations) | 1 | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 1
Abscess (Infections and infestations) | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1
Cystitis (Infections and infestations) | 1 | 0 | 0
Endophthalmitis (Infections and infestations) | 0 | 0 | 1
Infected Skin Ulcer (Infections and infestations) | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 1
Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0
Staphylococcal Sepsis (Infections and infestations) | 0 | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 1
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0
Wound Abscess (Infections and infestations) | 0 | 0 | 1
Wound Infection Staphlyococcal (Infections and infestations) | 0 | 0 | 1
Renal Failure Chronic (Renal and urinary disorders) | 1 | 1 | 6
Renal Failure (Renal and urinary disorders) | 1 | 0 | 2
Azotaemia (Renal and urinary disorders) | 1 | 0 | 1
Nephrotic Syndrome (Renal and urinary disorders) | 1 | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 1 | 0 | 1
Renal Impairment (Renal and urinary disorders) | 0 | 0 | 2
Cystitis Glandularis (Renal and urinary disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Renal Artery Stenosis (Renal and urinary disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 5
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 3 | 1
Diabetic foot (Metabolism and nutrition disorders) | 1 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 0
Fluid Retention (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Tibia Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Cervical Vertebral Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ligament Rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Multiple Injuries (Injury, poisoning and procedural complications) | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pelvic Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Perirenal Haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Renal Haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Spinal Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Upper Limb Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Burkitt's Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Laryngeal Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung Carcinoma Cell Type Unspecified Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Multiple Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Neuroendocrine Carcinoma of the Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Small Cell Lung Cancer Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Duodenal Ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Duodenal Ulcer Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Duodenitis (Gastrointestinal disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Entercolitis (Gastrointestinal disorders) | 0 | 1 | 0
Gastric Ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatic Disorder (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Umbilical Hernia, Obstructive (Gastrointestinal disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 3
Cerebral Ischaemia (Nervous system disorders) | 0 | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 0 | 1
Hypoglycaemic Coma (Nervous system disorders) | 0 | 0 | 1
Hypotonia (Nervous system disorders) | 0 | 0 | 1
Loss of Consciousness (Nervous system disorders) | 1 | 0 | 0
Orthostatic Intolerance (Nervous system disorders) | 1 | 0 | 0
Vertebrobasilar Insufficiency (Nervous system disorders) | 0 | 0 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 3
Aortic Stenosis (Vascular disorders) | 1 | 0 | 1
Circulatory Collapse (Vascular disorders) | 0 | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 1 | 0
Hypertensive Crisis (Vascular disorders) | 0 | 1 | 0
Peripheral Arterial Occlusive Disease (Vascular disorders) | 0 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 1
Nephrogenic Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Chest Pain (General disorders) | 1 | 1 | 0
Device Failure (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1
Hernia Obstructive (General disorders) | 0 | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 0 | 0 | 1
Diabetic Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Drug Eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Haemoglobin Decreased (Investigations) | 0 | 1 | 0
International Normalised Ratio Increased (Investigations) | 0 | 0 | 1
Drug Hypersensitivity (Immune system disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FCM (High Ferritin Target) (N=154) | FCM (Low Ferritin Target) (N=150) | Oral Iron (N=312)
Diarrhoea (Gastrointestinal disorders) | 15 | 11 | 45
Constipation (Gastrointestinal disorders) | 2 | 5 | 37
Nausea (Gastrointestinal disorders) | 9 | 7 | 15
Dyspepsia (Gastrointestinal disorders) | 2 | 3 | 17
Urinary Tract Infection (Infections and infestations) | 18 | 10 | 17
Nasopharyngitis (Infections and infestations) | 13 | 10 | 16
Influenza (Infections and infestations) | 4 | 8 | 7
Oedema Peripheral (General disorders) | 21 | 21 | 29
Back Pain (Musculoskeletal and connective tissue disorders) | 15 | 12 | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 7 | 15
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2 | 8 | 15
Hypertension (Vascular disorders) | 21 | 14 | 32
Hypotension (Vascular disorders) | 8 | 4 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 11 | 11
Dizziness (Nervous system disorders) | 9 | 8 | 7
Headache (Nervous system disorders) | 6 | 10 | 7
Anaemia (Blood and lymphatic system disorders) | 7 | 8 | 10

LIMITATIONS AND CAVEATS:
Initially 1,016 subjects were planned, but due to slow enrollment only 626 were randomised which was sufficient to make the primary comparison between FCM targeting high ferritin level and oral iron.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators may not present or publish partial or complete study results individually. Any manuscript or abstract proposed by the Investigators must be reviewed and approved in writing by Vifor Pharma before submission for publication. Names of all Investigators participating in the study will be included in the publication.